CLINICAL TRIAL: NCT00022282
Title: Neovastat (AE-941) in Refractory and Early Relapse Multiple Myeloma Patients
Brief Title: AE-941 in Treating Patients With Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AEterna Zentaris (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068801; AETERNA-AE-MM-00-02
Record Dates: First submitted 2001-08-10; First posted 2003-10-15 (Estimated); Last update posted 2013-02-28 (Estimated); Status verified 2008-02

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: refractory multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — shark cartilage extract

INTERVENTIONS:
Drug: shark cartilage extract AE-941

SUMMARY:
RATIONALE: AE-941 may help to slow the growth of multiple myeloma.

PURPOSE: Phase II trial to study the effectiveness of neovastat in treating patients who have relapsed or refractory multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the confirmed tumor response rate in patients with early relapse or refractory multiple myeloma treated with AE-941 (Neovastat).
* Determine the safety of this drug in these patients.
* Evaluate the time to progression in patients treated with this drug.
* Evaluate the duration of tumor response (partial response, response, and complete response) in patients treated with this drug.

OUTLINE: This is a multicenter, open-label study.

Patients receive oral AE-941 (Neovastat) twice daily.

Patients are followed every 4 weeks until disease progression.

PROJECTED ACCRUAL: A total of 125 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of multiple myeloma (MM) according to the Durie and Salmon criteria
* Refractory to or in early relapse after standard chemotherapy with or without stem cell transplantation
* Measurable disease

  * Quantifiable IgM, IgG, or IgA paraprotein in serum AND/OR
  * Bence-Jones protein in urine
* No plasma cell leukemia (more than 20% plasma cells in peripheral blood and an absolute plasma cell count of at least 2,000/mm3)
* No nonsecretory MM
* No spinal cord compression

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* More than 6 months

Hematopoietic:

* No clinical symptoms of hyperviscosity

Hepatic:

* Not specified

Renal:

* Creatinine no greater than 2 times upper limit of normal
* Calcium no greater than 11 mg/dL

Other:

* No other prior malignancy within the past 5 years except basal cell carcinoma of the skin or carcinoma in situ of the cervix
* No severe allergy to fish or seafood
* No medical condition that would interfere with intake and/or absorption of study medication (e.g., gastrectomy or major intestinal resection)
* No significant medical or psychiatric condition that would preclude study participation
* Not pregnant
* Negative pregnancy test
* Fertile patients must use adequate contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics
* No prior history of treatment with thalidomide for more than 14 days duration
* At least 4 weeks since prior biological therapy for MM
* Concurrent epoetin alfa allowed

Chemotherapy:

* See Disease Characteristics
* At least 4 weeks since prior chemotherapy for MM

Endocrine therapy:

* At least 4 weeks since prior steroid therapy for MM
* No prednisone maintenance therapy

Radiotherapy:

* At least 4 weeks since prior radiotherapy
* No concurrent palliative or curative radiotherapy

Surgery:

* Not specified

Other:

* At least 28 days since other prior shark cartilage products
* At least 28 days since other prior experimental therapeutic agents
* Concurrent monthly bisphosphonate (pamidronates) infusions allowed
* No other concurrent anticancer treatment
* No other concurrent shark cartilage products
* No other concurrent therapies for MM

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-04; Primary Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Québec, Canada